CLINICAL TRIAL: NCT03976739
Title: Study on the Effect of Bile Reflux on Gastric Cancer and Its Precancerous Lesions: a Multiple Center, Cross-sectional Study.
Brief Title: Study on the Effect of Bile Reflux on Gastric Cancer and Its Precancerous Lesions: a Cross-sectional Study.
Status: Completed | Type: Observational
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, Principal Investigator, Clinical Professor, Xijing Hospital of Digestive Diseases
Other Study IDs: KY20191026-F-1
Record Dates: First submitted 2019-05-27; First posted 2019-06-06 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2019-05

CONDITIONS: Bile Reflux Gastritis; Gastric Cancer; Helicobacter Pylori Infection; Intestinal Metaplasia; Precancerous Lesions
Keywords: gastric cancer; helicobacter pylori; precancerous lesion; bile reflux
MeSH Terms: conditions — Stomach Neoplasms; Bile Reflux

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- chronic gastritis: patients with chronic non-atrophic gastritis and chronic atrophic gastritis according to histopathological results
- precancerous lesion: patients with gastric intestinal metaplasia and intraepithelial neoplasia according to histopathological results
- gastric cancer: patients with gastric cancer according to histopathological results

SUMMARY:
To explore the effects of bile reflux on gastric cancer and its precancerous lesions, so as to better prevent the occurrence and development of gastric cancer.

DETAILED DESCRIPTION:
This study was a multicenter cross-sectional study. Patients were consecutively enrolled and divided into gastric cancer group, gastric precancerous lesions group, and chronic gastritis group, according to histopathological results. The bile reflux detection rate and Helicobacter pylori infection status were recorded for each group.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years old, gender is not limited;
2. patients with upper abdominal pain, abdominal distension, belching, anorexia, early satiety, hiccup, acid reflux, upper abdomen burning sensation and other upper gastrointestinal symptoms;
3. Voluntary acceptance of Hp testing;
4. Voluntary acceptance of the endoscopy and pathological biopsy.

Exclusion Criteria:

1. had undergone upper gastrointestinal surgery;
2. Previous diagnosis of esophageal cancer;
3. Previous diagnosis of gastric cancer;
4. Previous diagnosis of MALT lymphoma;
5. pregnant and lactating women;
6. Those with mental disorders;
7. Refusal to sign the informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients are from several centers all around the China
Sampling Method: Non-Probability Sample
Enrollment: 1162 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
corelation between the bile reflux and gastric mucosa diseases | up to 6 months
  we evaluate the corelation between the bile reflux and gastric mucosa diseases according to the histopathological results and the scales the patients finished

SECONDARY OUTCOMES:
the risk factors of primary bile reflux gastritis | up to 6 months
  we evaluate the the risk factors of primary bile reflux gastritis according to the scales and endoscopical results

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hosipital of Digestive Disease, Xi'an, Shaanxi, China